CLINICAL TRIAL: NCT05569538
Title: Phase 2 Study to Assess the Safety and Efficacy of Bomedemstat (IMG-7289) in Combination With Ruxolitinib in Patients With Myelofibrosis
Brief Title: Bomedemstat (IMG-7289) Plus Ruxolitinib for Myelofibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMG-7289-IIS001
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-10

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Bomedemstat; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Patients refractory to, relapsed or intolerant of ruxolitinib): (Experimental): Bomedemstat : The starting dose of bomedemstat at Initial Treatment Period Cycle 1 Day 1 will be 0.4 mg/kg daily for all patients in Cohort A. The first up-titration is not permitted until Initial Treatment Period Cycle 2 Day 1; thereafter, the dose may be up-titrated no more frequently than every 4 weeks from the prior up- or down-titration (note: down-titrations may occur at any time (or the current dose maintained) in the best interest and safety of the patient), to a target platelet count range of 50-100 x 10^9/L.
  Ruxolitinib: Patients will continue their prior, stable dose of ruxolitinib. This same dose will be continued throughout the study unless dose modification is required because of toxicity.
  Interventions: Drug: Bomedemstat
- Cohort B (Cohort B will consist of 10 patients who are JAK inhibitor naïve): (Experimental): Bomedemstat: The starting dose of bomedemstat at Initial Treatment Period Cycle 1 Day 1 will be 0.4 mg/kg daily for all patients in Cohort B. The first up-titration is not permitted until Initial Treatment Period Cycle 2 Day 1; thereafter, the dose may be up-titrated no more frequently than every 4 weeks from the prior up- or down-titration (note: down-titrations may occur at any time (or the current dose maintained) in the best interest and safety of the patient), to a target platelet count range of 50-100 x 10^9/L.
  Ruxolitinib: Patients will start treatment with ruxolitinib at Initial Treatment Period Cycle 1 Day 1. The starting dose of ruxolitinib will be 10 mg BID. This same dose will be continued throughout the study unless dose modification is required because of toxicity.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Bomedemstat will be self-administered orally once daily. In both cohorts, the dose of bomedemstat will be adjusted in each patient based on titration of the patient's platelet count to the target range. Ruxolitinib will be self-administered orally. Both medications will continue uninterrupted in 28-day cycles. Subjects will continue combination treatment through the Initial Treatment Period (first 6 cycles), which includes a Qualification Assessment. Those deriving clinical benefit in the opinion of the treating physician may continue receiving combination treatment in the Additional Treatment Period (6 cycles). Qualification Assessments will be performed at the end of each Additional Treatment Period, which is iterative, and may repeat for as long as clinical benefit is sustained, at the discretion of the treating physician.
  Other Names: IMG-7289

SUMMARY:
This is an open-label, Phase 2 study of bomedemstat (IMG-7289), an inhibitor of lysine-specific demethylase 1 (LSD1), in combination with JAK inhibition (JAKi) in patients with myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

1. Patients refractory to, relapsed or intolerant of ruxolitinib as per one of the below:

* Refractory is defined as <30% reduction in spleen length or <10% SVR compared to baseline having received ruxolitinib for ≥12 weeks prior to enrollment, AND on a stable dose for ≥8 weeks prior to starting investigational therapy
* Relapsed is defined as an increase in spleen volume of ≥25% by MRI/CT from nadir, or, ≥100% in palpable spleen length from a baseline of 5 to 10 cm BLCM or, ≥50% increase in spleen length from a baseline spleen length ≥10 cm BLCM
* Intolerance is defined as the development in patients treated with ruxolitinib for ≥28 days of:

  * Red blood cell transfusion requirement of 2 units/month for 2 months
  * Grade 3 thrombocytopenia, anemia, hematoma, and/or hemorrhage while on ruxolitinib treatment

Cohort B:

1. Patients who are JAK inhibitor naïve, AND:

   * Require MF-directed treatment, AND
   * Have measurable disease burden including one of the following:

     * Disease-related symptoms, determined by a MFSAF or MPN-SAF TSS of ≥10, or at least 2 symptoms with scores ≥3
     * Documented splenomegaly by physical exam, with spleen palpated ≥5 cm below the left costal margin

   Both Cohorts A and B:
2. Willing and able to provide informed consent
3. Age ≥18 years
4. Diagnosis of Overt Myelofibrosis (primary, post-ET, or post-PV) per World Health Organization (WHO) diagnostic criteria
5. Intermediate-1, Intermediate-2, or high-risk disease by Dynamic International Prognostic Scoring System (DIPSS)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Platelet count ≥100 x 10^9/L prior to dosing on Cycle 1 Day 1
8. Absolute neutrophil count ≥0.5 x 10^9/L prior to dosing on Cycle 1 Day 1
9. Peripheral blast count ≤10% prior to dosing on Cycle 1 Day 1
10. Able to swallow capsules
11. Women of childbearing potential and fertile men must agree to use an approved method of contraception from Screening until 30 days after the last dose of bomedemstat and ruxolitinib.

Exclusion Criteria:

1. Those with increased risk of bleeding, including any of the following:

   1. Activated partial thromboplastin time (aPTT) ≥1.3 x the local upper limit of normal
   2. International normalized ratio (INR) ≥1.3 x the local upper limit of normal
   3. Known history of a platelet function disorder
   4. Other known bleeding disorder that is active at the time of screening (Von Willebrand's disease, dysfibrinogenemia, hemophilia, etc.)
2. History of splenectomy or prior splenic irradiation
3. Use of an investigational agent within 14 days of study treatment (or at least 7 half-lives of that agent, whichever is longer), prior to the first dose of bomedemstat
4. Current use of monoamine oxidase A and B inhibitors (MAOIs)
5. Uncontrolled, active infection
6. Major surgery within 4 weeks of starting the study drug, or not recovered from side effects of surgery
7. Any other serious medical conditions that could compromise study participation, in the opinion of the investigator
8. Known HIV infection or known, active hepatitis B or hepatitis C infection
9. Concurrent second active and non-stable malignancy (patients with a concurrent second active but stable malignancy, i.e., non-melanoma skin cancers, are eligible)
10. Current use of a prohibited medication (e.g., romiplostim) or expected to require any of these medications during treatment
11. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to bomedemstat or LSD1 inhibitors (i.e., monoamine oxidase inhibitors; MAOIs) that contraindicates participation
12. Evidence at the time of Screening of significant renal or hepatic insufficiency (unless due to hemolysis) as defined by any of the following local lab parameters:

    1. Calculated glomerular filtration rate (GFR; using the Cockcroft-Gault equation) <40 mL/min or serum creatinine >1.5 x the local upper limit of normal
    2. Aspartate transaminase (AST) or alanine aminotransferase (ALT) ≥2.5 x the local upper limit of normal
13. Pregnant or lactating females, or females planning to become pregnant at any time during the study
14. Unwilling or unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 24 months
  Enumeration and description of adverse events (AEs), including determination of dose limiting toxicities (DLTs), serious adverse events (SAEs), and other AEs

SECONDARY OUTCOMES:
Spleen response at 24 weeks | 24 weeks
  Proportion of patients who experience a spleen length reduction by palpation of ≥30% OR spleen volume reduction (SVR) of ≥35% by MRI or CT by 24 weeks of treatment
Symptom response at 24 weeks | 24 weeks
  Proportion of patients who describe a ≥50% reduction in symptom burden by the Myelofibrosis Symptom Assessment Form (MFSAF) by 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — Department of Medicine, the University of Hong Kong
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No